CLINICAL TRIAL: NCT07137780
Title: Lokomat® Versus RoboGait®: Comparative Effects on Walking, Mobility, and Quality of Life Under Different Guidance Force Settings in Motor-Incomplete Spinal Cord Injury
Brief Title: Lokomat® vs RoboGait® Under Different Guidance Force Settings in Motor-Incomplete SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-MSS-03
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Robot-Assisted Gait Training; Functional Mobility; Guidance Force
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lok90- (GF < 90% with Lokomat®) (Experimental): Participants in this arm received robotic-assisted gait training using the Lokomat® V6 system (Hocoma AG, Switzerland) with an average guidance force (GF) of less than 90%. Training was conducted three times per week for 4 weeks, totaling 10 sessions. In addition to robotic gait training, participants also received conventional physiotherapy, including stretching, strengthening, balance, walking, and mobility exercises.
  Interventions: Device: Lokomat® V6 (GF < 90%)
- Lok90+ (GF ≥ 90% with Lokomat®) (Experimental): Participants in this arm received robotic-assisted gait training using the Lokomat® V6 system (Hocoma AG, Switzerland) with an average guidance force (GF) of 90% or higher. Training was conducted three times per week for 4 weeks, totaling 10 sessions. In addition to robotic gait training, participants also received conventional physiotherapy, including stretching, strengthening, balance, walking, and mobility exercises.
  Interventions: Device: Lokomat® V6 (GF ≥ 90%)
- RG (RoboGait®) (Experimental): Participants in this arm received robotic-assisted gait training using the RoboGait® system (BAMA Teknoloji, Türkiye) with an average guidance force (GF) of 90% or higher. Training was conducted three times per week for 4 weeks, totaling 10 sessions. In addition to robotic gait training, participants also received conventional physiotherapy, including stretching, strengthening, balance, walking, and mobility exercises.
  Interventions: Device: RoboGait®

INTERVENTIONS:
Device: Lokomat® V6 (GF < 90%) — Robotic-assisted gait training using the Lokomat® V6 system (Hocoma AG, Switzerland) with an average guidance force of less than 90%. Training was delivered three times per week for 4 weeks, totaling 10 sessions. In addition to robotic gait training, participants received conventional physiotherapy, including stretching, strengthening, balance, walking, and mobility exercises.
  Arms: Lok90- (GF < 90% with Lokomat®)
Device: Lokomat® V6 (GF ≥ 90%) — Robotic-assisted gait training using the Lokomat® V6 system (Hocoma AG, Switzerland) with an average guidance force of 90% or higher. Training was delivered three times per week for 4 weeks, totaling 10 sessions. In addition to robotic gait training, participants received conventional physiotherapy, including stretching, strengthening, balance, walking, and mobility exercises.
  Arms: Lok90+ (GF ≥ 90% with Lokomat®)
Device: RoboGait® — Robotic-assisted gait training using the RoboGait® system (BAMA Teknoloji, Türkiye) with an average guidance force of 90% or higher. Training was delivered three times per week for 4 weeks, totaling 10 sessions. In addition to robotic gait training, participants received conventional physiotherapy, including stretching, strengthening, balance, walking, and mobility exercises.
  Arms: RG (RoboGait®)

SUMMARY:
This study compares two robotic-assisted gait training systems, Lokomat® and RoboGait®, used under different guidance force (GF) settings, in people with motor-incomplete spinal cord injury (iSCI). Nineteen adults, aged 18 years or older, with injury at T3 level or below and classified as AIS C or D within two years of injury, participated. They were assigned to one of three groups based on the average GF used during training: Lok90- (GF < 90% with Lokomat®), Lok90+ (GF ≥ 90% with Lokomat®), and RG (GF ≥ 90% with RoboGait®). All participants completed 10 treadmill-based gait training sessions over 4 weeks, in addition to standard physiotherapy including stretching, strengthening, balance, and walking exercises. Walking ability, mobility, muscle strength, balance, independence in daily activities, and quality of life were assessed before and after the program. The study aimed to see whether the type of robot and GF setting affected recovery. Results showed modest improvements in some outcomes, with changes depending on the group and outcome measured. Findings suggest that adjusting GF settings may help tailor robotic gait training to individual needs.

DETAILED DESCRIPTION:
This pilot study investigated the effects of two robotic-assisted gait training systems, Lokomat® V6 (Hocoma AG, Switzerland) and RoboGait® (BAMA Teknoloji, Türkiye), applied under different guidance force (GF) settings, on walking ability, functional mobility, and health-related quality of life in individuals with motor-incomplete spinal cord injury (iSCI).

Eligible participants were aged 18 years or older, with injury at T3 level or below, AIS C or D classification, and injury duration of 2 years or less. Exclusion criteria included severe spasticity (Modified Ashworth Scale ≥ 3), joint disorders, implanted electronic devices, orthostatic hypotension, cardiac problems, or conditions preventing secure positioning in the robotic systems.

Participants were assigned to three groups according to their average GF during training: Lok90- (GF < 90% with Lokomat®), Lok90+ (GF ≥ 90% with Lokomat®), and RG (GF ≥ 90% with RoboGait®). All participants completed 10 treadmill-based gait training sessions over 4 weeks, with three sessions per week. Walking speed and angular parameters were individually adjusted to enhance comfort, reduce fatigue, and encourage active participation. Alongside robotic gait training, all participants received conventional physiotherapy that included stretching, strengthening, balance, walking, and mobility exercises.

The primary outcome was walking status, measured using the Walking Index for Spinal Cord Injury II (WISCI II). Secondary outcomes included, functional mobility (Timed Up and Go Test, TUG), lower extremity muscle strength (LEMS), balance (Berg Balance Scale, BBS), functional independence (Spinal Cord Independence Measure III, SCIM III), and health-related quality of life (WHOQOL-BREF-TR). The study aimed to determine whether the type of robotic system and GF settings influence functional outcomes in iSCI rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosis of spinal cord injury (SCI) at T3 level or below.
* Injury duration of no more than 2 years.
* Functional classification of C or D based on the American Spinal Injury Association (ASIA) Impairment Scale.
* ICD-10 diagnosis codes between S24.73-S24.77 or S34.70

Exclusion Criteria:

* Participation in another study.
* Joint disorders affecting mobility.
* Implanted electronic devices.
* Orthostatic hypotension.
* Severe spasticity in the lower extremities (Modified Ashworth Scale score ≥ 3).
* Cardiac problems or conditions impairing stabilization in the robotic systems.
* Presence of a colostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-11-23 (Actual)

PRIMARY OUTCOMES:
Walking Index in Spinal Cord Injury II | 24 months
  Walking Index in Spinal Cord Injury II for walking independence level assessment

SECONDARY OUTCOMES:
Timed Up and Go Test | 24 months
  Timed Up and Go Test overground walking assessment
Berg Balance Scale | 24 months
  Berg Balance Scale for balance assessment
ASIA Lower Extremity Muscle Score | 24 months
  Assessment of lower extremity muscle strength using the American Spinal Injury Association (ASIA) Lower Extremity Motor Score (LEMS)
Spinal Cord Independence Measure (SCIM III) | 24 months
  Spinal Cord Independence Measure (SCIM III) for activity of daily living assessment
World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) | 24 months
  World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) for quality of life assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)